CLINICAL TRIAL: NCT03532230
Title: Prospective, Multi-center, Cohort Study of the Cost Effectiveness of Osteopathic Manipulative Treatment for Chronic Low Back Pain
Brief Title: Cost Effectiveness of OMT for Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Rowan University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Richard Jermyn, DO, Director of the NeuroMusculoskeletal Institute (NMI) and Professor and Chair of Rehabilitation Medicine, Rowan University
Other Study IDs: AOA-OMT
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Lumbar Radiculopathy; Lesion of Sciatic Nerve, Left Lower Limb; Lesion of Sciatic Nerve, Right Lower Limb; Lumbar Spinal Stenosis; Lumbar Spondylosis; Lumbago With Sciatica, Left Side; Lumbago With Sciatica, Right Side
Keywords: Chronic Low Back Pain; Osteopathic Manipulative Medicine
MeSH Terms: conditions — Radiculopathy; Sciatic Neuropathy; Spinal Stenosis; Spondylosis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: 90 new patients seeking treatment for chronic low back pain. This group will receive standard care plus osteopathic manipulative treatment (OMT) for low back pain.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- Control Group: 90 new patients seeking treatment for chronic low back pain. This group will receive only standard care without osteopathic manipulative treatment (OMT) for low back pain.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — No specific OMT techniques will be required for the present study. However, data on the number of OMT sessions patients receive will be collected.
  Groups: Experimental Group

SUMMARY:
The specific aim of this study is to conduct a prospective, multicenter cohort study over four months to compare the cost of standard of allopathic care (control group, N=90) versus standard of care plus osteopathic manipulative treatment (experimental group, N=90) in a cohort of 180 consecutive patients seeking treatment for chronic low back pain at three osteopathic clinics and three allopathic medical clinics (offering only standard care) located in three different regions of the United States.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic low back pain (lasting more than 3 months) who are between 18 to 84 years old will be eligible for the study. Inclusion criteria will be specified by the following the 2017/2018 International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes associated with chronic low back pain:
* M54.16 Lumbar radiculopathy
* G57.01 Lesion of sciatic nerve, right lower limb
* G57.02 Lesion of sciatic nerve, left lower limb
* M48.061 Lumbar spinal stenosis, without neurogenic claudication
* M48.062 Lumbar spinal stenosis, with neurogenic claudication
* M47.816 Lumbar spondylosis
* M48.07 Lumbar spinal stenosis, lumbosacral
* M54.41 Lumbago with sciatica, right side
* M54.42 Lumbago with sciatica, left side

Exclusion Criteria:

* Patients with diabetic neuropathy, congenital lumbar and sacral abnormalities, lumbar fracture, multiple myeloma, metastatic bone disease, history of spinal and/or pain lasting less than three months will be excluded from the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, multicenter, observational study will follow two groups of patients over four months. The first (experimental) group will be 90 new patients seeking treatment for chronic back pain at three osteopathic clinics. The experimental group will receive standard of care plus osteopathic manipulative treatment (OMT) for low back pain.
  The second (control) group will be 90 new patients who will receive only standard care without OMT for chronic low back pain as delivered at a local pain clinic.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Total Costs | 4 months
  The cost data will be collected from the electronic medical record of each patient enrolled in the study. Because the costs for comparable treatments vary with respect to different socioeconomic and geographic regions in the United States, the mean total-healthcare costs per patient will be calculated based on codes for 2018 Medicare fee schedules for each clinic listed in the Current Procedural Terminology (CPT) for office visits, medications, OMT, and referrals.

SECONDARY OUTCOMES:
Total Morphine-Equivalents | 4 months
  Various pain medications that might have been prescribed will be calculated and compared to morphine equivalents at admission to the study and after four months at each of the treatment centers.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jermyn, DO, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (3):
- United States (3):
  - Michigan State University, East Lansing, Michigan
  - Rowan University SOM NeuroMusculoskeletal Institute, Stratford, New Jersey
  - The Pain Associates, Voorhees Township, New Jersey